CLINICAL TRIAL: NCT06387615
Title: Evaluating the Impact of Non-Invasive Brain Stimulation on Learning and Consolidation of Phonologically Similar Novel Spoken Words
Brief Title: Impact of Non-invasive Brain Stimulation on Learning Novel Spoken Words
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, C. Nikki Arrington, PhD, Assistant Research Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H22086; 1R21HD108576-01A1 (NIH)
Record Dates: First submitted 2024-04-11; First posted 2024-04-29 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Dyslexia; Dyslexia, Developmental; Learning; Developmental Disorder, Reading
Keywords: word learning; consolidation; vocabulary; artificial lexicon; brain stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Dyslexia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active cTBS (Experimental): Active cTBS will be administered to the left supramarginal gyrus
  Interventions: Other: Active cTBS
- Sham stimulation (Sham Comparator): Sham stimulation will be administered to the left supramarginal gyrus
  Interventions: Other: Sham

INTERVENTIONS:
Other: Active cTBS — Active stimulation
  Arms: Active cTBS
Other: Sham — Control stimulation
  Arms: Sham stimulation

SUMMARY:
The purpose of the proposed study is to use transcranial magnetic stimulation (TMS) to evaluate a neurobiological model of spoken word learning in older youth. Specifically, it is hypothesized that: (1) inhibition of the left dorsal stream will impact subsequent learning, processing, and retention of phonologically similar pseudowords; (2) the impact of dorsal stream inhibition on word learning will be associated with baseline levels of variability in neural activity, indicative of underlying differences in cortical excitability.

DETAILED DESCRIPTION:
The proposed study is designed to assess the contribution of the dorsal stream of the language network (i.e., left supramarginal gyrus, or SMG) to different aspects of novel word learning in two groups of participants (16-24 years of age): 20 typically developing older youth (OYTD; tested in Aim 1) and 20 older youth with reading difficulties (OYRD; tested in Aim 2). The investigators will use inhibitory continuous theta burst stimulation (cTBS), a well-established repetitive TMS (rTMS) protocol that reduces cortical excitability in a targeted brain region for up to 60 minutes. Participants will complete a baseline magnetic resonance imaging (MRI) session in Week 1, followed by cTBS or sham stimulation to the left SMG, with order of administration counterbalanced across participants. Immediately following cTBS (or sham), participants will complete a visual pseudoword phonological discrimination task and a spoken word learning task. The following day (i.e., 24 hours later), retention of items learned will be measured. In Week 2, cTBS (or sham) will be administered to the left SMG (whichever stimulation was not administered in Week 1) and then the pseudoword discrimination and word learning tasks will be administered using a different set of novel words from those presented in Week 1. Twenty-four hours later, the retention of this second set of items will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Native English speaker (who is not fluent in any other language and does not identify as bilingual)
* Normal or corrected to normal vision

Exclusion Criteria:

* Diagnosed with Autism Spectrum Disorder
* Hearing deficits (>25 decibels at 500+ Hz), visual deficits (>20/40), serious emotional problems (e.g., severe, uncontrolled depression) and certain neurological conditions (e.g., uncontrolled seizure disorders)
* Individuals with certain metals in their bodies or with certain health conditions. If an individual has braces on their teeth, a cardiac pacemaker; hearing aid; other metal in their body or eyes (which may include certain metallic-embedded tattoos), including but not limited to pins, screws, shrapnel, plates, dentures or other metal objects
* Individuals taking certain medications that lower seizure threshold
* Individuals with TMS Screening and Contraindication Forms which do not pass TMS Tech review
* Individuals with MRI Screening and Contraindication Forms which do not pass MRI Tech review

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Novel Word Learning Task | 5-mins post stimulation; 24hrs post stimulation
  The spoken word learning task, completed post-cTBS, will consist of a two-alternative forced choice paradigm in which participants will be presented with two pictures of unusual objects, and will be asked to indicate via button press which picture matches a spoken label. Initial trials require a pure guess, with feedback provided on each trial, and continued until a correct answer is given. Across six learning blocks (24 trials each), participants will learn a set of eight pseudowords total. Twenty-four hours following the initial learning task, participants will be asked to complete two additional learning blocks which will be used to assess retention accuracy. Over the course of the experiment, participants will learn two different sets of items, counter-balanced across participants and groups.
Pseudoword Discrimination Task | Immediately following cTBS
  The visual pseudoword discrimination task is a computerized forced-choice, reaction time assessment of phonological processing. It measures the participants' ability to phonetically decode a string of letters. This task is simple with high accuracy and has proven highly sensitive to individual differences in phonological decoding skills. Participants are asked to judge via button press whether a visually presented letter string can be pronounced like a 'real word' or not.

SECONDARY OUTCOMES:
MRI Scan | baseline
  Pre-rTMS MRI scans will consist of anatomical and functional sequences consistent with well-established protocols in the field designed to assess baseline properties and functioning of the reading and language network. The functional MRI (fMRI) Picture Identification task is simple with high accuracy and has proven highly sensitive to individual differences in reading skills. Participants are asked to indicate via button press whether a target stimulus (written or spoken word) matches a picture cue. The fMRI Fast Localizer task rapidly presents sets of four words that vary based on orthographic, phonological, or semantic properties. Anatomical scans are necessary for localizing brain regions targeted for cTBS.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia State University/Georgia Tech Center for Advanced Brain Imaging (CABI), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The Open Science Framework (OSF) will be engaged to facilitate research integration in multiple aspects including collaboration among personnel, study design, data collection and analyses, and publication access. In addition, neuroimaging and behavioral data will be shared by depositing it in the Collaborative Informatics and Neuroimaging Suite (COINS), a platform hosted by Georgia State University/Georgia Institute of Technology/Emory University Center for Translational Research in Neuroimaging and Data Science (TReNDS). TReNDS allows for safe and secure data sharing with external users without granting access to protected health information. For preprints, platforms such as PsyArXiv and OSF Preprints will be used based on appropriate content area. All personnel will commit to use OSF to publicly share evaluation and research components.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Timely submission of raw data to repositories will provide an additional layer of safety. Neuroimaging data will be uploaded to COINS in real time. Cleaned behavioral datasets will be uploaded to OSF biannually. Metadata, code, small datasets and links to large datasets used in publications will be archived as supplements or on OSF. Publication specific data will be deposited to the OpenNeuro platform upon publication. All shareable data from this project will be made publicly available no later than the end of the project period, and any data associated with a publication will be made available at the time of publication. The latest point at which data will be provided to the archive is when articles using that data are accepted for publication, or at the conclusion of the project (whichever comes first).
Access Criteria: Any physical data for this project will be stored within locked filing cabinets for print copies and digital files will be encrypted and stored on password-protected secure servers separately from any participant code keys. Archived data will be stored on a secure server at Georgia State University when primary planned analyses of the data have been completed. The server will be backed up regularly using a tape backup system. The partition where data will sit on the server will not be accessible to anyone outside of the team.
  Audit trails are maintained for each file to document changes and deletions, and older versions of files are retrievable in the event of unintentional modification.

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Olson R, Forsberg H, Wise B, Rack J. Measurement of word recognition, orthographic, and phonological skills. In: Frames of Reference for the Assessment of Learning Disabilities: New Views on Measurement Issues. Paul H. Brookes Publishing Co.; 1994:243-277.